CLINICAL TRIAL: NCT03294213
Title: Prospective Non-interventional Evaluation of Intubation and Intensive Care Use of the New aScope™ 4 Broncho and aView
Status: Completed | Type: Observational
Sponsor: Ambu A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: CIS-002
Record Dates: First submitted 2017-09-22; First posted 2017-09-26 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Bronchoscopy; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- aScope 4 Broncho: The only data to be obtained are evaluation forms directly related to the users' perception of the aScope™ 4 Broncho
  Interventions: Device: aScope 4 Broncho

INTERVENTIONS:
Device: aScope 4 Broncho — Investigator is asked: "In your memory, compare your daily bronchoscope and the aScope 4 Broncho just evaluated" on patients admitted to the OR or ICU undergoing at least one bronchoscopy procedure Patients will not be asked to consent to participate in this study, as no patient data are obtained and the CE-marked aScope™ 4 Broncho is used within its intended use

SUMMARY:
This study is designed as a prospective observational, non-controlled, non-interventional study.

The aim of this study is to obtain a broad user perspective of the aScope™ 4 Broncho, focusing on the device functionalities within regular clinical practice and therapeutic use of flexible bronchoscopes in the OR and ICU.

The study will include a minimum of 100 adult patients admitted to the operating room (OR) or Intensive Care Unit (ICU) undergoing at least one bronchoscopy procedure. The inclusion will stop when 100 fully evaluable patients or a maximum of 150 patients have been enrolled.

The involved sites will include patients during a five months' period, from September 2017 to January 2018.

DETAILED DESCRIPTION:
Refer to brief description

ELIGIBILITY:
Inclusion Criteria:

* Patient's ≥18 years
* Clinical indication and eligible for an airway procedure involving a bronchoscopy procedure, as judged by the Investigator
* Patients being admitted in the OR or ICU at the investigational site

Exclusion Criteria:

- None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient's ≥18 years, Clinical indication and eligible for an airway procedure involving a bronchoscopy procedure, as judged by the Investigator, Patients being admitted in the OR or ICU at the investigational site
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pia Nordmand, MSc, Study Chair — Ambu A/S
Locations (1):
- Klinik für Anästhesiologie, Universitätsmedizin Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | aScope 4 Broncho
Started | 176
Completed | 176
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | aScope 4 Broncho
Number analyzed (Participants) | 176
Age, Continuous [Mean (Full Range); unit: years] — Population: Age Data were not collected
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex/Gender data were not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 60
  Denmark | 35
  Sweden | 14
  United Kingdom | 67

OUTCOME MEASURES:

1. Primary Outcome: User Preference of Scope
Description: This non-interventional study compared the clinical performance of the Ambu aScope 4TM Bron-cho with the standard bronchoscope (reusable or single-use) normally used at each of the study centers based on the investigators memory of the standard bronchoscope.
Time Frame: Data on patients from September 2017 to January 2018, investigators memory assessed immediately following use of the aSCope 4TM Broncho at each patient visit
Measure: Count of Participants; unit: Participants
Arm/Group | aScope 4 Broncho
Number analyzed (Participants) | 175
Participants
  Prefer aScope 4 Broncho | 103
  Prefer standard bronchoscope | 37
  No preference on bronchoscope | 35

ADVERSE EVENTS:
Time Frame: Data collected over the course of 5 months, Adverse Events assessed during each procedure
Arm/Group | aScope 4 Broncho
All-Cause Mortality (participants affected / at risk) | 0/176
Serious Adverse Events (participants affected / at risk) | 0/176
Other Adverse Events (participants affected / at risk) | 2/176
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | aScope 4 Broncho (N=176)
Poor light (Product Issues) | 1
Freezing image and blackout for 60 seconds (Product Issues) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT03294213/Prot_SAP_000.pdf